CLINICAL TRIAL: NCT03740334
Title: Phase I Trial of Ribociclib in Combination With Everolimus and Dexamethasone in Children and Young Adults With Relapsed Acute Lymphoblastic Leukemia
Brief Title: Ribociclib in Combination With Everolimus and Dexamethasone in Relapsed ALL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Andrew E. Place, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-328
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia ALL
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ribociclib; Dexamethasone; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ribociclib (RIBO) + Dexamethasone (DEX) (Experimental): * Ribociclib administered daily for 21 consecutive days
  * Dexamethasone administered intravenously on days 1-5 and again on days 11-15
  Interventions: Drug: Ribociclib; Drug: Dexamethasone
- RIBO + Everolimus (EVE) + DEX (Experimental): * Ribociclib administered daily for 21 consecutive days
  * Dexamethasone administered intravenously on days 1-5 and again on days 11-15
  * Everolimus administered daily for 21 consecutive days
  Interventions: Drug: Ribociclib; Drug: Dexamethasone; Drug: Everolimus
- RIBO + EVE+ DEX (dose expansion) (Experimental): * Ribociclib administered daily for 21 consecutive days. Dosing at RDE
  * Dexamethasone administered intravenously on days 1-5 and again on days 11-15
  * Everolimus administered daily for 21 consecutive days. Dosing at RDE
  Interventions: Drug: Ribociclib; Drug: Dexamethasone; Drug: Everolimus

INTERVENTIONS:
Drug: Ribociclib — Ribociclib, blocks a specific type of protein called a cyclin-dependent kinases (CDK)
  Other Names: LEE011
Drug: Dexamethasone — Corticosteroids are commonly used to treat ALL.
Drug: Everolimus — Everolimus is an inhibitor of mTOR. mTOR inhibition blocks the translation of genes that regulate cancer cell proliferation
  Other Names: Zortress
  Arms: RIBO + EVE+ DEX (dose expansion); RIBO + Everolimus (EVE) + DEX

SUMMARY:
This research study is evaluating a drug called ribociclib (LEE011) given in combination with everolimus and other standard of care chemotherapy drugs as a possible treatment for relapsed or refractory ALL.

The names of the drugs involved in this study are:

* ribociclib
* everolimus
* dexamethasone

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug or a combination of drugs. Phase I studies try to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug and the combination of drugs are still being studied.

The FDA (the U.S. Food and Drug Administration) has not approved the study drugs, ribociclib or everolimus, for relapsed ALL, but these drugs have been approved for other uses.

Ribociclib is a chemotherapy drug that is approved by the FDA for the treatment of certain types of breast cancer. It has also been studied in children and adults with other types of cancer. Information from these research studies has suggested that ribociclib may also be effective in treating participants with leukemia that did not respond to standard treatment or participants with leukemia that has come back after standard treatment.

The growth and survival of leukemia cells is controlled by proteins within the cancer cell. The study drug, ribociclib, blocks a specific type of protein called a cyclin-dependent kinases (CDK). Laboratory and other studies suggest that when ribociclib blocks CDKs, cancer cells stop growing.

Everolimus is a chemotherapy drug that is approved by the FDA for the treatment of breast cancer, neuroendocrine tumor and kidney cancer. Laboratory and other studies suggest that everolimus may prevent leukemia cell growth and also that it has been shown to increase the effectiveness of other chemotherapy drugs, including ribociclib. It has been studied in hundreds of people with various types of cancer as a single agent (a drug that is used alone to treat the cancer) or in combination with a number of other drugs.

The drug combination of ribociclib and everolimus has not been previously tested in children, though these agents have been used together in adults with breast cancer.

In this research study the investigators are looking to learn more about how ribociclib and everolimus work in combination with other standard of care drugs commonly used to treat relapsed/refractory leukemia. The main goals of the study are:

* To evaluate the side effects (good and/or bad) of giving ribociclib in combination with other standard of care drugs.
* To determine the highest dose of ribociclib and everolimus that can be given safely in combination with other standard of care drugs.
* To determine the amount of ribociclib and everolimus in the blood when it is given in combination with other standard of care drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 months (365 days) and ≤ 30 years
* Histologically confirmed diagnosis of either 1) relapsed or refractory ALL or 2) CML in lymphoid blast crisis (must have failed at least 2 lines of TKI therapy)

  * Primary refractory disease: Persistent disease after at least two induction attempts
  * Relapsed disease: Second or subsequent relapse, or any relapse refractory to salvage chemotherapy
* Participants must have bone marrow with ≥ 1% lymphoblasts definitively identified either on a bone marrow aspirate or biopsy sample, as assessed by morphology, immunohistochemical studies, flow cytometry, karyotype, cytogenetic testing such as fluorescent in situ hybridization (FISH) or other molecular studies.
* Participants with CNS1 or CNS2 disease are eligible. Patients with isolated CNS relapse or CNS 3 disease are not eligible. (Refer to Section 12.4 for definitions of CNS status)
* Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study and meet all of the following criteria:
* Corticosteroids: 14 days must have elapsed since the completion of systemic corticosteroid administration. The following uses of corticosteroids are permitted: single doses (e.g., during anesthesia), topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airway diseases, asthma), eye drops or local injections (e.g., intra-articular)
* Myelosuppressive chemotherapy: 14 days must have elapsed since the completion of myelosuppressive therapy. Individuals may have received any of the following medications within 14 days without a "wash-out" period:

  * Standard maintenance therapy, other than corticosteroids (vincristine, 6MP, low dose methotrexate)
  * Hydroxyurea
  * Intrathecal chemotherapy with methotrexate, hydrocortisone and/or cytarabine.
* Radiation therapy (XRT):

  * Total Body Irradiation (TBI) or cranial radiation therapy: Must have been completed more than 90 days prior to study entry
  * XRT for chloroma does not require a washout period.
  * Palliative XRT does not require a washout
* Small molecule inhibitors (BCR-ABL or FLT3 inhibitors, for example): 7 days must have elapsed since the completion of therapy. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair.
* Immunotherapy: At least 6 weeks after the administration of any type of immunotherapy, including, but not limited to, tumor vaccines, chimeric antigen receptor (CAR) therapy, other immune effector cell therapy or checkpoint inhibitors.
* Monoclonal antibodies: At least 3 half-lives of the antibody after the last dose of a monoclonal antibody. (See table on DVL homepage listing monoclonal antibody half-lives: https://members.childrensoncologygroup).
* Prior hematopoietic stem cell transplant (HSCT): Patients who have received HSCT are eligible, but must meet all of the following conditions:

  * Autologous HSCT > 60 days of study entry
  * Allogeneic HSCT > 90 days of study entry
  * No evidence of graft-versus-host-disease (GVHD)
  * Weaning or stable doses of calcineurin inhibitors are permitted provided there is no evidence of active GVHD.
* Participants must have a body surface area (BSA) ≥ 0.4 m2.
* Performance status:

  --Lansky > 50 for individuals < 16 years old; Karnofsky > 50% for individuals ≥ 16 years old (See Appendix A).
* Participants must have adequate organ function as defined by the following laboratory values:

  * Direct bilirubin ≤1.5 X institutional upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) < 3 x ULN for age and aspartate aminotransferase (AST) < 3 x ULN for age. Patients with leukemic infiltration of the liver must have AST and ALT < 5 x ULN for age.
  * Creatinine below institutional ULN or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Echocardiogram ejection fraction ≥50%. Echocardiogram must be obtained while patient is not receiving cardiotropic medications (e.g., pressors or afterload reducers).
* QTcF < 450 ms on screening ECG.
* Oxygen saturation ≥ 90% by pulse oximetry without administration of supplemental oxygen.
* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 21 days after the last dose of the study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, documented using an institutionally approved informed consent procedure.

Exclusion Criteria:

* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of ribociclib, everolimus or dexamethasone (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Individuals with CNS 3 leukemia at time of study entry. History of CNS 3 disease is allowable as long as patient meets eligibility criteria (CNS 1 or 2) at time of enrollment.
* Individuals with Down syndrome.
* Treatment with hematopoietic growth factors (G-CSF):

  * Long-acting (e.g., Neulasta) within 14 days prior to study entry
  * Short-acting (e.g., Neupogen) within 7 days prior to study entry
* Treatment with an investigational agent within 28 days of study entry, or 3 half-lives, whichever is longer.
* Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Cardiomyopathy
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
* Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

  * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure or history of significant/symptomatic bradycardia.
  * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication (See Appendix C for list of prohibited medications)
  * Inability to determine the QTcF interval on screening EKG (using Fridericia's correction)
* Prior exposure to a CDK4/6 inhibitor
* Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug (see Appendix C for prohibited medications):

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * Medications with a narrow therapeutic window that are predominantly metabolized through CYP3A4/5
  * Herbal preparations/medications, dietary supplements.
* Patients refractory to red blood cell or platelet transfusions.
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Patients with systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment.
* Patients known to have human immunodeficiency virus (HIV) infection; baseline testing for HIV is not required.
* Patients known to have active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen); baseline testing for viral hepatitis is not required.
* Major surgery within 2 weeks of the first dose of study drugs. The following are not considered major surgery for the purposes of eligibility: Tumor biopsy, insertion of a gastric feeding tube, central venous access.
* Individuals with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Individuals with a history of a different malignancy (other than ALL) are ineligible except for the following circumstances:

  * Individuals are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy.
  * Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Pregnant or nursing women are excluded

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic analysis - AUC(0-24hr): | 3 years
  Blood samples obtained for Pharmacokinetic (PK) analysis will be used to describe how study drugs are distributed and metabolized by human subjects. Samples for PK analysis will be obtained during Cycle 1 of all Cohorts. Area under the concentration-time curve from time zero to 24 hours (AUC(0-24hr)) is a measure of a subject's exposure to study drugs.
Pharmacokinetic analysis - Cmax | 3 years
  Blood samples obtained for Pharmacokinetic (PK) analysis will be used to describe how study drugs are distributed and metabolized by human subjects. Samples for PK analysis will be obtained during Cycle 1 of all Cohorts. Maximum observed concentration (Cmax) will be determined from the plasma concentration data
Pharmacokinetic analysis - Tmax | 3 years
  Blood samples obtained for Pharmacokinetic (PK) analysis will be used to describe how study drugs are distributed and metabolized by human subjects. Samples for PK analysis will be obtained during Cycle 1 of all Cohorts. Time of first observation of Cmax (tmax) will be determined from the plasma concentration data
Toxicity assessments | 3 years
  Toxicities experience by study subjects will be reported and graded for severity using CTCAE version 5. These data will contribute to determining the Maximum tolerated dose (MTD)
Maximum Tolerated Dose (MTD) | 3 years
  This dose, determined by review of toxicity data, will define the highest dose that is tolerable in this patient population.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 3 years
  Preliminary anti-leukemic activity of the combinations of ribociclib, everolimus and dexamethasone will be reported. Bone marrow and cerebrospinal fluid evaluations will occur at the end of each cycle. ORR will be defined as the number of patient experiencing complete remission (CR), complete remission with incomplete platelet recovery (CRp), complete remission with incomplete count recovery (CRi) and partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Place, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor-Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor-Investigator or designee].